CLINICAL TRIAL: NCT02452775
Title: A Randomized Pilot Trial to Test the Addition of Montanide and Polyiclc to Autologous Oxidized Tumor Cell Lysate Vaccine in Combination With Gmcsf in Primary Advanced Epithelial Ovarian, Primary Peritoneal, or Fallopian Tube Cancer
Brief Title: Autologous OC-L Vaccine and Ovarian Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: Ovarian Cancer Research Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 40814
Record Dates: First submitted 2015-05-21; First posted 2015-05-25 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Primary Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms | interventions — Monatide (IMS 3015); poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (4):
- Arm 1 (Experimental): Subjects in ARM 1 will receive the vaccination with OC-L alone
  Interventions: Biological: OC-L
- Arm 2 (Experimental): subjects in ARM 2 will receive vaccination with OC-L admixed with Montanide,
  Interventions: Other: Montanide
- Arm 3 (Experimental): subjects in ARM3 will receive vaccination with OC-L admixed with 1 mg poly-ICLC (Hiltonol)
  Interventions: Other: poly-ICLC (Hiltonol),
- Arm 4 (Experimental): subjects in ARM 4 will receive vaccination with OC-L admixed with both Montanide and 1 mg poly-ICLC.
  Interventions: Biological: OC-L; Other: Montanide; Other: poly-ICLC (Hiltonol),

INTERVENTIONS:
Biological: OC-L
  Arms: Arm 1; Arm 4
Other: Montanide
  Arms: Arm 2; Arm 4
Other: poly-ICLC (Hiltonol),
  Arms: Arm 3; Arm 4

SUMMARY:
This is a randomized pilot trial to test the addition of 2 investigational agents, Montanide and poly-ICLC (a TLR3 agonist) to a backbone of autologous oxidized tumor cell lysate vaccine (OC-L) administered with GMCSF in subjects with primary epithelial ovarian, fallopian tube, or primary peritoneal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has primary ovarian (including low malignant potential), fallopian tube, or primary peritoneal cancer FIGO stage III or IV defined surgically at the completion of initial abdominal surgery.
2. Subject has had cytoreductive surgery and has completed first line platinum based chemotherapy in an adjuvant or neo-adjuvant setting as part of standard of care treatment.
3. Subject has no evidence of disease based on radiographical imaging
4. Subject has appropriate tissue available from the cytoreductive surgery tumor lysate preparation.
5. Lysate must meet release criteria.
6. Subject is 18 years of age or older.
7. Subject has an ECOG performance status of ≤ 2.
8. Subject understood and signed the study specific informed consent.
9. Subjects screened between 1 to 12 weeks after last cycle of chemotherapy.
10. Subjects screened any time after completed last cycle of chemotherapy till progression or first recurrence of the disease.
11. Subject has had at least 4 weeks of postoperative recovery from surgery prior to enrollment to ensure complete wound healing.
12. Subjects who screen fails can be re-enrolled if the causation of the screen fail has been corrected.

Exclusion Criteria:

1. Subject for whom tumor lysate does not meet release criteria
2. Subject has a positive serum Yo antibody (Does not need to be repeated if performed in the past)
3. Subject has a chronic or acute hepatitis C infection. Subject with an old infection that has cleared may be included.
4. Subject has a chronic or acute hepatitis B infection. Subject with an old infection that has cleared may be included.
5. Subject has positive test result at the screening visit for one or more of the following:

   1. HTLV-1/2
   2. Anti-HIV 1 Antibody (α-HIV-1)
6. Subject requires or is likely to require more than a two-week course of corticosteroids for intercurrent illness. Subject must complete the course of corticosteroids 2 weeks before screening to meet eligibility.
7. Subject has renal insufficiency as defined by a serum creatinine > 2.2 mg/dl or BUN > 40 mg/dl. Note: If creatinine is greater than 1.5 x ULN, creatinine clearance must be greater than 60ml/min.
8. Subject has proteinuria > 3.5 gm over 24 hrs are not eligible for the study
9. Subject with liver failure as defined by a serum total bilirubin > 2.0 and/or serum transaminases > 3X the upper limits of normal.
10. Subject has hematopoietic failure at baseline as defined by one of the following:

    1. Platelets < 100,000/ mm3
    2. WBC < 2,500/mm3
    3. Absolute Neutrophil Count (ANC) < 1,000/mm3
    4. Absolute lymphocyte count < 200/ mm3
    5. Hematocrit < 30%
11. Subject has any acute infection that requires specific therapy. Acute therapy must have been completed within seven days prior to study enrollment.
12. Subject has a serious, non-healing wound, ulcer, or bone fracture.
13. Subject has a clinically significant cardiovascular disease including:

    1. Uncontrolled hypertension;
    2. Myocardial infarction or unstable angina within 6 months prior to enrollment
    3. New York Heart Association (NYHA) Grade II or greater congestive heart failure
14. Subject has a grade II or greater peripheral vascular disease.
15. Subject has a clinically significant peripheral artery disease, e.g., those with claudication, within 6 months.
16. Subject has any underlying conditions, which would contraindicate therapy with study treatment
17. Subject has organ allografts.
18. Subject is receiving medication(s) that might affect immune function. Use of H2 antagonists are prohibited as are all antihistamines five days before and five days after each injection of study vaccine. However, NSAIDS including COX-2 inhibitors, acetaminophen or aspirin are permitted.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Numbers of Adverse Events | 3.5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Ovarian Cancer Research Center, Philadelphia, Pennsylvania, United States